CLINICAL TRIAL: NCT03666780
Title: Lifetech LAmbre™ Left Atrial Appendage (LAA) Closure System Post-Market Clinical Follow-up: MULTI-CENTER, SINGLE-ARM, PROSPECTIVE, POST-MARKET STUDY
Brief Title: Lifetech LAmbre™ Left Atrial Appendage (LAA) Closure System Post-Market Clinical Follow-up Study
Acronym: LISA
Status: Completed | Type: Observational
Sponsor: Lifetech Scientific (Shenzhen) Co., Ltd. (Industry)
Collaborators: IQVIA Biotech (Industry)
Responsible Party: Sponsor
Other Study IDs: LA-PMCF-01
Record Dates: First submitted 2018-09-10; First posted 2018-09-12 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Atrial Fibrillation
Keywords: Left Atrial Appendage Occluder; LAmbre; Lifetech LAA; Lifetech LAmbre; LT LAA; Left Atrial Appendage
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subject: All patients who signed informed consent and are implanted with a Lifetech LAmbre occluder device will undergo follow-up (FU) evaluations as per local hospital standards and corresponding IFU which is expected to be at the following time points post-implant:
  * At discharge (+/- 1 day)
  * 1-3 months (+/- 1 week)
  * 6 months (+/- 2 weeks)
  * 12 months (+/- 1 month)
  * 2 years (+/- 3 month)
  * 3 years(+/- 3 month)
  Patients who have undergone a LAmbre explant should remain in the study and adhere to the above-mentioned follow-up time point until completion of 3-year follow-up period.
  After the patient has completed the 3-year follow-up assessments, the patient is considered to have completed the study. A study exit eCRF needs to be completed and the patient will receive routine care.
  Interventions: Device: LAmbre Occluder

INTERVENTIONS:
Device: LAmbre Occluder — All patients are implanted with Lifetech LAmbre occluder device.

SUMMARY:
Multi-center, single-arm, prospective, post-market study of LAmbre™ LAA Closure System. To evaluate the immediate and long-term procedural success of Lifetech LAmbre™ occluders in patients.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common cardiac arrhythmia causing ischemic stroke. The CHA2DS2-VASc score was developed to estimate the stroke rate in patients with non-valvular AF, and high scores predict a raised annual stroke risk. The yearly stroke risks without treatment in patients with CHA2DS2-VASc Scores 2 and 9 are 2.2% and 15.2% respectively. For patients with increased stroke risk (CHA2DS2-VASc score ≧2), warfarin or other novel oral anticoagulants (NOAC) are recommended for stroke prevention.

Despite the effectiveness of current pharmacological therapies for stroke prevention in atrial fibrillation, around 20% of patients discontinue therapy - whether new oral anticoagulants (NOAC) or warfarin because of side effects and/or bleeding. In addition, warfarin needs to be dosed individually to target an international normalized ratio (INR) of 2-3 for striking an optimal balance between bleeding and ischemic stroke events. This, combined with drug-drug interaction that occurs with both NOACs and warfarin, results in inadequate stroke protection in a substantial portion of AF patients. The LAA is the source of 90% of cardiac emboli attributed to stroke events. This is a windsock-like structure on the lateral border of the left atrium with internal trabeculations, and being a confined space is prone to blood stasis and thrombus formation.

Currently, there are surgical, epicardial, and percutaneous techniques for occluding this structure in order to reduce stroke in AF patients who cannot take long-term oral anticoagulants, and the percutaneous route is intuitively the most attractive given its relative non-invasiveness. The two devices in most widespread use for percutaneous LAA closure worldwide are the Watchman (Boston Scientific, Natick, MA, USA) and the Amplatzer Cardiac Plug (ACP) (Abbott, IL, CA USA). However, both devices have limitations including the need for relatively large delivery sheaths (9-14 French) and limited recapture and repositioning capabilities.

LAmbre™ LAA Closure System (Lifetech Scientific, Shenzhen, China) is a novel self-expanding LAA occluder constructed from a nitinol mesh and polyester membranes and consists of an umbrella and a cover connected by a short central waist. The device is delivered by an 8-10 French sheath and has full recapture and repositioning capabilities. LAmbre™ LAA Closure System received the CE mark in June 2016.

This PMCF study will be carried out following the CE mark of the LAmbre™ LAA Closure System and is intended to confirm the effectiveness and safety of the LAmbre™ LAA Closure System.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be at least 18 years of age;
2. Patients with non-valvular paroxysmal, persistent, or permanent atrial fibrillation with long-term sustainability scheduled for interventional LAA closure;
3. Patient characteristics consistent with the corresponding IFU and sizing guidelines*;

   * Note: Choose a device that is 3-8mm larger than the landing zone diameter.
4. The patient or legally authorized representative has been informed of the nature of the study, agrees to its provisions, and has provided written informed consent, approved by the appropriate Ethics Committee (EC);
5. The patient agrees to comply with the requirements of the study including the 3-year follow-up.

Warning: The device sizing is based on angiographic measurements.

Exclusion Criteria:

1. Any contra-indication mentioned in the corresponding IFU*;

   * Note: In IFU, the Left Atrial Appendage Closure System is contraindicated for the following:

     1. Patients' LAA anatomy is not suitable for the REF of the device.
     2. Patients with intracardiac thrombus.
     3. Patients with active endocarditis or other infections causing bacteremia.
     4. Patients where the placement of the device would interfere with any intracardiac or intravascular structures.
     5. Patients with contraindications to X-ray and/or trans-esophageal echocardiographic examinations.
     6. Patients with known hypersensitivity to nickel.
2. Currently participating in other investigational drug- or device studies;
3. Patient who is pregnant, planning to become pregnant or breastfeeding;
4. Patients cannot tolerate transoesophageal echocardiogram (TEE).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with non-valvular paroxysmal, persistent, or permanent atrial fibrillation with long-term sustainability are scheduled for interventional LAA closure.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2018-11-16 (Actual); Primary Completion 2021-11-29 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Absence of peri-procedural stroke/TIA, device embolization, cardiac or vascular perforation, any other device or procedure-related serious adverse event or death (procedure or device-related or of unknown cause); | Within 7 days post-procedure.
  Peri-procedure defined as within 7 days of the procedure.
Implant success. | At procedure.
  Implant success is defined as the correct positioning and release of the occluder device into the proper anatomical location. Correct positioning is assessed as the absence of major residual jet flow (>5mm) into the LAA closure with the device evaluated by the transesophageal echocardiogram (TEE).

SECONDARY OUTCOMES:
Incidence of stroke or systemic embolism or death through 3 years post-implantation. | From attempted procedure to 3 years post-implantation
  Incidence of stroke or systemic embolism or death through 3 years post-implantation.
Successful sealing around the device at the LAA orifice with residual jet ≤5 mm flow measured by TEE at 1-3 months, 6 months post-implantation. | 1-3 months, 6 months post-implantation
  Successful sealing around the device at the LAA orifice with residual jet ≤5 mm flow measured by TEE at 1-3 months, 6 months post-implantation.
Device or procedure-related Serious Adverse Events (SAEs) from attempted procedure through 3 years post-implantation | From attempted procedure to 3 years post-implantation
  Device or procedure-related Serious Adverse Events (SAEs) from attempted procedure through 3 years post-implantation.
All SAEs (death included) from attempted procedure through 3 years post-implantation. | From attempted procedure to 3 years post-implantation
  All SAEs (death included) from attempted procedure through 3 years post-implantation.

CONTACTS AND LOCATIONS:
Overall Officials: Horst Sievert, Prof, Principal Investigator — CVC CardioVasculäres Centrum Frankfurt
Locations (26):
- 1001 - HKU Queen Mary Hospital, Hong Kong, China
- 201 - Aarhus Universitetshospital, Aarhus, Denmark
- Germany (13):
  - 104 - Charité Campus Benjamin Franklin (CBF), Berlin
  - 107 - Charité Campus Virchow-Klinikum, Berlin
  - 105 - UKB Universitätsklinikum Bonn, Bonn
  - 111 - Klinikum Coburg GmbH, Coburg
  - 114 - Facharztzentrum Dresden-Neustadt GbR, Dresden
  - 102 - Alfried Krupp Hospital Ruettenscheid, Essen
  - 101 - CVC CardioVasculäres Centrum Frankfurt, Frankfurt
  - 109 - Cardioangiologisches Centrum Bethanien (CCB), Frankfurt
  - 108 - Universitätsklinikum Jena, Jena
  - 103 - Klinikum St. Georg gGmbH, Leipzig
  - 110 - Herzzentrum Leipzig (HZL), Leipzig
  - 113 - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - 106 - Peter Osypka Herzzentrum, München
- 301 - Mater Misericordiae University Hospital, Dublin, Ireland
- Italy (4):
  - 401 - Centro Cardiologico Monzino, Milan
  - 403 - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - 406 - Clinica Mediterranea S.P.A./Clinica Mediterranea - Ospedale e Centro Diagnostico, Napoli
  - 405 - La Struttura ASL Roma 2, Roma
- 501 - Wojewódzki Specjalistyczny Szpital im. dr. Wł. Biegańskiego, Lodz, Poland
- Spain (3):
  - 603 - FundacióInstitut Hospital del Mar d'Investigacions Mèdiques (IMIM), Barcelona
  - 602 - Hospital Clínic de Barcelona, Barcelona
  - 601 - University Hospital of Salamanca/Hospital Clínico Universitario de Salamanca, Salamanca
- 801 - Sahlgrenska Universitetssjukhuset/Sahlgrenska University Hospital, Gothenburg, Sweden
- 901 - Faculty of Medicine Ramathibodi Hospital, Mahidol University, Bangkok, Thailand